CLINICAL TRIAL: NCT03072472
Title: BowelScope: Accuracy of Detection Using ENdocuff Optimisation of Mucosal Abnormalities
Acronym: B-ADENOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Collaborators: ARC Medical Design Ltd (Unknown); Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-ADENOMA
Record Dates: First submitted 2017-01-16; First posted 2017-03-07 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Neoplasms; Colonic Polyp; Adenoma; Neoplasia GI; Digestive System Neoplasms; Intestinal Neoplasms; Neoplasms, Glandular and Epithelial; Digestive Disease; Intestinal Diseases; Colonic Diseases; Rectal Diseases; Intestinal Polyps; Polyps; Pathological Conditions, Anatomical
Keywords: Colorectal Cancer; Endoscopy; Screening; Colonic Adenoma; Adenoma Detection Rate; Endocuff; Endocuff Vision
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps; Adenoma; Digestive System Neoplasms; Intestinal Neoplasms; Neoplasms, Glandular and Epithelial; Digestive System Diseases; Intestinal Diseases; Colonic Diseases; Rectal Diseases; Intestinal Polyps; Polyps; Pathological Conditions, Anatomical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocuff-assisted Flexible Sigmoidoscopy (Experimental): Patients in this arm will receive their screening sigmoidoscopy with the Endocuff Vision in situ on the scope
  Interventions: Device: Endocuff Vision
- Standard Flexible Sigmoidoscopy (No Intervention): Patients in this arm will receive their screening sigmoidoscopy without the Endocuff on the scope

INTERVENTIONS:
Device: Endocuff Vision — The EndocuffTM (ARC Medical Design Ltd and Diagmed, UK) is a device (CE marked in UK) made of a soft plastic material with a unique dynamic shape. Endocuff Vision™ is placed snugly around the colonoscope tip prior to insertion. It does not project beyond the tip of the scope, providing an unrestricted view. It helps anchor the scope tip against the bowel wall to provide a stable platform of access. The soft, elastic projections are pushed back (recoiled) towards the scope shaft during insertion but evert during withdrawal to hold colon folds away from the field of view.
  Arms: Endocuff-assisted Flexible Sigmoidoscopy

SUMMARY:
This study aims to assess the effect, if any, on the adenoma detection rate of BowelScope bowel cancer screening flexible sigmoidoscopies by using the Endocuff Vision device.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the fourth most common cancer in the UK with 40,000 new cases diagnosed annually. Most CRCs arise from the adenoma-carcinoma sequence which is a process that can take up to 10 years. Population screening programmes allow for earlier detection and removal of adenomas that may become malignant over time thus reducing CRC mortality. The English Bowel Scope Screening (BSS) programme began in 2013 and invites adults aged 55 and above for a one-off flexible sigmoidoscopy. The aim of the BSS programme is to reduce CRC development via the adenoma-carcinoma sequence through the detection and removal of adenomas from the left side of the colon. A large UK study has shown that offering one-off flexible sigmoidoscopy screening with adenoma clearance to adults aged 55-64 years reduced CRC incidence by 23% and mortality by 31%. Adenoma detection rate (ADR) is the most important marker of mucosal visualisation and is a surrogate marker of high quality colonoscopy. Data from colonoscopy studies have illustrated that a 1% increase in ADR is associated with a 3% decrease in interval colorectal cancer. In the BSS programme, ADR is comparatively lower the that shown in the initial sigmoidoscopy screening trials with a wide variation between endoscopists. Another marker that is often used is adenoma miss rates which also demonstrate a wide variation in clinical practice. Reasons for lesions not being detected at flexible sigmoidoscopy can be extrapolated from colonoscopy data and include; suboptimal technique; shorter withdrawal time; inadequate bowel preparation; presence of flat, depressed or subtle lesions; and the inability to visualise the proximal side of haustral folds, flexures (blind spots) and rectal valves. With the aid of the colonoscopic cuff Endocuff Vision®, the investigators aim to improve visualisation of the colonic mucosa by flattening colonic folds and manipulating them away from the field of forward view the investigators hypothesise that the Endocuff Vision® will improve adenoma detection rates by providing better fold retraction, a wider field of view and better scope tip stabilisation. This clinical randomised study will be conducted in subjects referred and scheduled for screening flexible sigmoidoscopy via the NHS English Bowel Scope Screening (BSS) Programme and will compare Endocuff Vision®-Assisted Flexible Sigmoidoscopy (EAFS) with Standard Flexible Sigmoidoscopy (SFS).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and over
2. Referral for screening flexible sigmoidoscopy
3. Ability to give informed consent

Exclusion Criteria:

1. Absolute contraindications to flexible sigmoidoscopy
2. Established or suspicion of large bowel obstruction or pseudo-obstruction
3. Known colon cancer or polyposis syndromes
4. Known colonic strictures
5. Known severe diverticular segment (that is likely to impede sigmoidoscope passage)
6. Patients with known active colitis (ulcerative colitis, Crohn's colitis, diverticulitis, infective colitis)
7. Patients lacking capacity to give informed consent
8. Patients who are on clopidogrel, warfarin, or other new generation anticoagulants which have not been stopped for the procedure as these will preclude polyp removal
9. Pregnancy

Ages: 55 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3221 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate | Day of procedure
  Proportion of examinations expressed as a percentage where at least one adenoma is found

SECONDARY OUTCOMES:
Mean adenomas detected per procedure | Day of procedure
  Number of adenomas found in each procedure
Rate of cuff exchange | Day of procedure
  How often the cuff is removed
Non-inferiority of complete withdrawal time in procedures where no polyps are detected | Day of procedure
  Length of procedure in minutes and seconds
Compare overall procedure time between groups | Day of procedure
  Length of procedure in minutes and seconds
Measure differences in ADR accounting for patient procedure based variables (e.g. accounting for extent of examination and bowel preparation). | Day of procedure
  Proportion of examinations expressed as a percentage where at least one adenoma is found
Compare the rate of discovered cancers between groups | On histology check 48-72 hours post procedure
  Number of cancers found
Examination extent between groups based on presumed anatomical location with a straight endoscope | Day of procedure
  Anatomical location
Examination extent between groups based on distance of insertion in centimetres with a straight endoscope | Day of procedure
  Depth of insertion in centimetres
Patient satisfaction between groups using the Gloucester scale of assessment of patient comfort | Day of procedure
  Numerical 4 point patient comfort score
Identify any difference in future colonoscopic workload produced by increased ADR in terms of number of patients referred for full colonoscopy between the EAFS and SFS groups. | Day of procedure
  Number of additional colonoscopies required
Compare the ADR of the first 20% of patients scoped by each colonoscopist with the last 20% of patients in each arm to identify any changes in ADR to assess any learning curve effect. | 18 months
  Proportion of examinations expressed as a percentage where at least one adenoma is found
Compare the baseline ADR of each colonoscopist prior to trial recruitment with their individual ADR in patients where EndocuffTM Vision was not used. | 18 months
  Proportion of examinations expressed as a percentage where at least one adenoma is found

CONTACTS AND LOCATIONS:
Overall Officials: Colin J Rees, MBBS MRCP FRCP, Principal Investigator — South Tyneside and Sunderland NHS Foundation Trust
Locations (16):
- United Kingdom (16):
  - South Tyneside NHS Foundation Trust, South Shields, Tyne and Wear
  - Bolton NHS Foundation Trust, Bolton
  - Gloucestershire Hospitals NHS Foundation Trust, Cheltenham
  - Dorset Healthcare University NHS Trust, Dorchester
  - County Durham and Darlington NHS Foundation Trust, Durham
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Kendal
  - Kettering General Hospital NHS Trust, Kettering
  - North West London Hospitals NHS Trust, London
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Oxford Health NHS Trust, Oxford
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Pennine Acute Hospitals NHS Trust, Rochdale
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - North Tees and Hartlepool NHS Trust, Stockton-on-Tees
  - West Hertfordshire Hospitals NHS Trust, Watford
  - The Royal Wolverhamptom NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rees CJ, Brand A, Ngu WS, Stokes C, Hoare Z, Totton N, Bhandari P, Sharp L, Bastable A, Rutter MD, Verma AM, Lee TJ, Walls M; B-ADENOMA trial group comprises. BowelScope: Accuracy of Detection Using Endocuff Optimisation of Mucosal Abnormalities (the B-ADENOMA Study): a multicentre, randomised controlled flexible sigmoidoscopy trial. Gut. 2020 Nov;69(11):1959-1965. doi: 10.1136/gutjnl-2019-319621. Epub 2020 Apr 3. PMID 32245908